CLINICAL TRIAL: NCT02005354
Title: Does Trans-Cutaneous Electrical Nerve Stimulation (TENS) Alleviate The Pain Experienced During Bone Marrow Sampling in Addition to Standard Techniques?A Randomised, Double-Blinded, Controlled Trial
Brief Title: Does Trans-Cutaneous Electrical Nerve Stimulation (TENS) Alleviate The Pain Experienced During Bone Marrow Sampling?
Acronym: TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: Torbay and South Devon NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13/P/168
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Pain
Keywords: Pain; Bone marrow aspiration; trephine biopsy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trans-cutaneous Electrical Nerve Stimulation (TENS) (Active Comparator): The Intervention-TENS group will have 2 electrodes applied proximal to the painful area along neuro-anatomical distribution (electrode-one placed 5cm superior and 2cm medial to the posterior superior iliac spine and electrode-two placed 5cm medial to the posterior superior iliac spine) in the same way as the control-TENS group.
  The concealed electrical parameter in this group will be within the therapeutic window, that is, well above the sensory detection threshold but below the pain threshold giving a "strong but comfortable sensation". From previous studies, this is likely to be 50-110Hz.
  The device will be activated prior to entry into the treatment room and 2 minutes before administration of local anaesthetic and for 2 minutes after removal of the biopsy needle. This will cover the expected duration of pain as assessed in the pilot study.
  All patients will receive standard pain relief (ie. local anaesthetic with or without inhaled nitrous oxide)
  Interventions: Device: Trans-cutaneous Electrical Nerve Stimulation (TENS); Drug: Standard pain relief (ie. local anaesthetic with or without inhaled nitrous oxide)
- Trans-cutaneous Electric Nerve Stimulation (TENS) (Placebo Comparator): Patients in the CT group will have 2 gel-electrodes applied proximal to the sampling area (usually the right posterior superior iliac crest).
  The Control-TENS device will be identical in appearance to the "Intervention-TENS" device with a functioning display panel. The concealed electrical parameter in this group will be titrated to and set at the sensory detection.
  All patients will receive standard pain relief (ie. local anaesthetic with or without inhaled nitrous oxide)
  Interventions: Device: Trans-cutaneous Electrical Nerve Stimulation (TENS); Drug: Standard pain relief (ie. local anaesthetic with or without inhaled nitrous oxide)

INTERVENTIONS:
Device: Trans-cutaneous Electrical Nerve Stimulation (TENS) — Patients in whom a bone marrow biopsy is planned will be randomised to one of two groups - a Placebo Comparator group where the TENS machine will be set at the lowest sensory threshold and an Active Comparator group where the TENS machine will be set at a recognised analgesic level (>50Hz and below the pain threshold for the patient).
Drug: Standard pain relief (ie. local anaesthetic with or without inhaled nitrous oxide) — All patients will receive standard pain relief (ie. local anaesthetic with or without inhaled nitrous oxide)

SUMMARY:
The approach of this study will be to answer the question does high-frequency stimulation Trans-Cutaneous Electrical Nerve Stimulation (TENS) alleviate the pain experienced during the bone marrow sampling procedure in addition to the standard analgesia given (ie. local anaesthetic with or without inhaled nitrous oxide).

Null hypothesis: TENS does not alleviate the pain experienced during the bone marrow sampling procedure in addition to the standard analgesia given

DETAILED DESCRIPTION:
Patients in whom a bone marrow biopsy is planned will be randomised to one of two groups - a control-TENS group where the TENS machine will be set at the lowest sensory threshold and an intervention-TENS group where the TENS machine will be set at a recognised analgesic level (>50 Hertz (Hz) and below the pain threshold for the patient) (Bennett et al. 2011). The identity of the TENS type will be concealed from both the patient and the doctor performing the biopsy. The primary outcome will be pain and this will be recorded by the patient immediately after the procedure using a validated numerical scale (0-10). All patients will receive standard pain relief (ie. local anaesthetic with or without inhaled nitrous oxide).

The benefit of this study is to establish whether or not TENS can benefit patients as an additional, safe, non-invasive and inexpensive method of pain relief during this frequently painful procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Participants are those medical patients seen in the haematology outpatients clinic for whom a bone-marrow trephine biopsy is deemed necessary either for diagnosis, staging or disease monitoring purposes. Participants are either new patients or routine follow ups.
* Participant is able (in the Investigators opinion) and willing to comply with all study requirements.
* Participant is willing to allow his or her General Practitioner to be notified of participation in the study.

Exclusion Criteria:

* Any known adverse reaction to high-frequency TENS or electrode gel pads
* Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon AJ Rule, MBChB, MPhil, Study Director — University Hospital Plymouth NHS Trust; Sarah L Poplar, MB ChB, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom

REFERENCES:
- [Background] Bennett MI, Hughes N, Johnson MI. Methodological quality in randomised controlled trials of transcutaneous electric nerve stimulation for pain: low fidelity may explain negative findings. Pain. 2011 Jun;152(6):1226-1232. doi: 10.1016/j.pain.2010.12.009. Epub 2011 Mar 23. PMID 21435786
- [Derived] Tucker DL, Rockett M, Hasan M, Poplar S, Rule SA. Does transcutaneous electrical nerve stimulation (TENS) alleviate the pain experienced during bone marrow sampling in addition to standard techniques? A randomised, double-blinded, controlled trial. J Clin Pathol. 2015 Jun;68(6):479-83. doi: 10.1136/jclinpath-2015-202908. Epub 2015 Mar 10. PMID 25759407

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 patients were randomised, thirty five patients received TENS impulses at a strong but comfortable amplitude (intervention group) and 35 patients received TENS impulses just above the sensory threshold (control group)
Groups:
- TENS Intervention: The concealed electrical parameter in this group will be within the therapeutic window, that is, well above the sensory detection threshold but below the pain threshold giving a "strong but comfortable sensation". From previous studies, this is likely to be 50-110Hz.
  The device will be activated prior to entry into the treatment room and 2 minutes before administration of local anaesthetic and for 2 minutes after removal of the biopsy needle. This will cover the expected duration of pain as assessed in the pilot study.
  All patients will receive standard pain relief (ie. local anaesthetic with or without inhaled nitrous oxide)
- TENS Placebo Comparator: Placebo Comparator group where the TENS machine will be set at the lowest sensory threshold and an Active Comparator group where the TENS machine will be set at a recognised analgesic level (>50Hz and below the pain threshold for the patient).
  Standard pain relief (ie. local anaesthetic with or without inhaled nitrous oxide): All patients will receive standard pain
Period: Overall Study
Arm/Group | TENS Intervention | TENS Placebo Comparator
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients were >18 years & required a bone marrow for diagnosis, staging or disease monitoring. Patients with known adverse reaction to TENS or electrode gel pads and patients with a cardiac pacemaker or implantable defibrillator in-situ were excluded from the trial. There was no upper age limit.
Groups:
- Total: Total of all reporting groups
Arm/Group | TENS Intervention | TENS Placebo Comparator | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Full Range); unit: years] | 68 [55 to 83] | 69 [41 to 86] | 69 [41 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Perception of Pain Will be Measured Using a Validated Numerical 0-10 Pain Scale Where 0 = no Pain and 10 = Worst Possible Pain
Description: To establish the effect of high-frequency stimulation TENS on the pain experienced by patients undergoing a bone-marrow biopsy, using standard technique with local anaesthetic.
  The perception of pain will be measured using a pain scale directly after and 24 hours after bone-marrow sampling in patients randomly allocated and blinded to the use of intervention-TENS (IT) or control-TENS (CT) in addition to local anaesthesia.
Time Frame: Post procedure and 24 hours
Measure: Mean (95% Confidence Interval); unit: Numerical Pain Severity Scale (0-10)
Arm/Group | TENS Intervention | TENS Placebo Comparator
Number analyzed (Participants) | 35 | 35
Numerical Pain Severity Scale (0-10)
  Mean Pain Score immediately post procedure | 5.6 [4.8 to 6.4] | 5.7 [4.8 to 6.6]
  Mean pain score 24 hours post procedure | 1.9 [1.2 to 2.6] | 1.9 [1.1 to 2.6]

ADVERSE EVENTS:
Time Frame: 11 months
Description: As per protocol
Arm/Group | TENS Intervention | TENS Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes